CLINICAL TRIAL: NCT03171766
Title: Pre-operative Neurocognitive Disorder and Low Near-infrared Spectrometry is Associated With Postoperative Delirium in Neurosurgical Patients
Brief Title: Pre-operative Neurocognitive Disorder and Low Near-infrared Spectrometry is Associated With Postoperative Delirium
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Hospitalar do Porto (Other)
Responsible Party: Principal Investigator, Pedro Amorim, MD, MD, Centro Hospitalar do Porto
Other Study IDs: 2016.253(216-DEFI/205-CES)
Record Dates: First submitted 2017-05-29; First posted 2017-05-31 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Neurocognitive Disorders; Postoperative Period; Postoperative Complications
MeSH Terms: conditions — Neurocognitive Disorders; Postoperative Complications | interventions — Visual Analog Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Mini-Mental State Examination (MMSE) — It is simple scored form of the cognitive mental status examination which includes eleven questions and requires only 5 to 10 minutes.
Diagnostic Test: Visual Analog Scale (VAS) — Visual Analog Scale (VAS) for pain score (including aphasia, motor disability, major neurocognitive disorder, etc)
Diagnostic Test: Mini Cog test — The Mini-Cog© test is another validated and simple tool to screen for dementia and cognitive dysfunction. It measures the cognitive reserve at the time of acute stress with a low degree of interobserver variability.

SUMMARY:
The main goal of the investigation is to identify the incidence of cognitive dysfunction and POD in patients older than 65 years of age undergoing neurosurgical elective surgery and determine if an association between cognitive dysfunction, basal NIRS and POD exists.

DETAILED DESCRIPTION:
Postoperative delirium (POD) is a common problem among elders who undergo surgery and anesthesia, with major health consequences. This investigation is expected to clarify and understand the role of neurocognitive reserve in the occurrence of POD, provide grounds to preoperative cognitive risk stratification and early preventive interventions to improve patients' outcomes. The surgical procedure and anesthesia are stressor events that interact with underlying risk factors and play an important role in the development of POD. Evidence is lacking to make recommendations on anesthesia related perioperative interventions. This investigation will contribute to better understand the association between types of anesthesia, medications, monitoring and other anesthesia related factors that can be a target for preventive interventions. This research will add knowledge and clarify the role of predictors and precipitant factors that might enlighten future research on risk stratification models and interventions, prognostic significance, and treatment implications for POD.

All patients scheduled for Neurosurgery will be approached the day before surgery to assess if inclusion criteria are met and obtain informed consent. If so, preoperative evaluation will be performed by two nurse investigators responsible for admission of patients in the Neurosurgical ward.

The Mini-Cog test and the will be administered before surgery to all participants as cognitive assessment tool. The social-economical status will be evaluated regarding the level of education in years, level of physical activity, occupation, income and number of languages spoken (all categorized with appropriate scales). Also, during the preoperative evaluation, demographic data, alcohol consumption, smoking, use of visual or hearing aids, comorbidities, usual medication and preoperative laboratory test results will be obtained and recorded in a form. On the day of the surgery, as the patient arrives at the Operating Room (OR), the anesthesiologist will check for informed consent and the patient will be monitored with the following with the standard ASA protocol.

The Near-infrared spectroscopy (NIRS) is a technology widely used in clinical investigation as an index of brain and tissue oxygenation. The INVOS© Cerebral/Somatic Oximetry is used in high-risk patients or surgeries to provide continuous, real-time, regional oxygen saturation (rSO2. The monitoring parameters, excluding the INVOS©, will be continuously recorded on the software program RugloopII© Waves (Demed, Genk, Belgium).

In the Post-Anesthesia Care Unit (PACU) the infrared pupillometer will be used to measure the patient pupillary reflexes 15 minutes after admission and before PACU discharge.

All included patients will be followed postoperatively from day 1 to the last day in-hospital, if hospitalized for less than 3 days, or until day 3. The investigator nurse will apply the Nu-DESC daily as a tool to screen delirium. The CAM will be applied to diagnose delirium if the patient is screened with POD. Pain will be evaluated using a standard 100mm VAS for pain (VAS=0 no pain, VAS=100 worst pain). Before hospital discharge all participants will retake the Mini-Cog test and the MMSE.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 65 years or older scheduled for elective Neurosurgery

Exclusion Criteria:

* refusal to give informed consent; inability to understand and cooperate to perform the Mini Cog test, Mini Mental State Examination (MMSE) and Visual Analog Scale (VAS) for pain score (including aphasia, motor disability, major neurocognitive disorder, etc); previous dementia documented on clinical records and Portuguese not first language.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 years or older scheduled for elective Neurosurgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-10-15 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
POD | From day 1 to the last day in-hospital, if hospitalized for less than 3 days, or until day 3.
  Incidence of Postoperative Disfunction

SECONDARY OUTCOMES:
Mortality | From day 1 to the last day in-hospital, if hospitalized for less than 3 days, or until day 3.
  Occurrence of In-hospital mortality
Complications | From day 1 to the last day in-hospital, if hospitalized for less than 3 days, or until day 3.
  Occurrence of Postoperative complications
Hospital length of stay | From day 1 to the last day in-hospital, if hospitalized for less than 3 days, or until day 3.
  Hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Susano, MD, Principal Investigator — Centro Hospitalar do Porto; Humberto Machado, PhD, Study Chair — Centro Hospitalar do Porto; Pedro Amorim, MD, Principal Investigator — Centro Hospitalar do Porto
Locations (1):
- Centro Hospitalar do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Susano MJ, Dias M, Seixas FS, Vide S, Grasfield R, Abelha FJ, Crosby G, Culley DJ, Amorim P. Association Among Preoperative Cognitive Performance, Regional Cerebral Oxygen Saturation, and Postoperative Delirium in Older Portuguese Patients. Anesth Analg. 2021 Mar 1;132(3):846-855. doi: 10.1213/ANE.0000000000005159. PMID 33002925